CLINICAL TRIAL: NCT02258906
Title: Effect of Ulinastatin on Postoperative Renal Function in Patients Undergoing Robot-assisted Laparoscopic Partial Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2014-0633
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Renal Mass
MeSH Terms: interventions — urinastatin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ulinastatin group (Experimental): Patients in the ulinastatin group are given ulinastatin during operation.
  Interventions: Drug: ulinastatin
- control group (Placebo Comparator): Patients in the control group receive the same volume of normal saline during operation.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: ulinastatin
  Arms: Ulinastatin group
Drug: normal saline
  Arms: control group

SUMMARY:
Ulinastatin reduces systemic inflammatory responses and protects organs from ischemia/reperfusion-induced injury. The aim of this study is to evaluate the effect of ulinastatin on postoperative renal function in patients undergoing robot-assisted laparoscopic partial nephrectomy. Seventy patients, aged 20 to 79 years, scheduled for robot-assisted laparoscopic partial nephrectomy will be divided into ulinastatin (n=35) and control (n=35) groups. Randomly selected patients of the ulinastatin group are given ulinastatin. In contrast, patients in the control group receive an equivalent volume of normal saline as a placebo. The primary endpoints are postoperative renal function measured by serum creatinine, cystatin C, and urine output.

ELIGIBILITY:
Inclusion Criteria:

* patients who are scheduled to undergo robot-assisted laparoscopic partial nephrectomy with an American Society of Anesthesiologists (ASA) physical status I-III

Exclusion Criteria:

* Subjects are ineligible if they have severe respiratory or cardiovascular disease, renal insufficiency before operation, cognitive dysfunction, are unable to communicate or speak Korean

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
postoperative renal function | for 3 days after surgery
  Postoperative renal function measured by serum creatinine, cystatin C, and urine output

SECONDARY OUTCOMES:
systemic inflammatory response | for 3 days after surgery
  the systemic inflammatory response measured by WBC, Neutrophil (%), and CRP

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea